CLINICAL TRIAL: NCT03012698
Title: Pilot Study for Testing Safety of Repetitive Magnetic Stimulation for Treatment of Dry Eye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epitech Mag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-10002
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Dry Eye; Sjogren's Syndrome; Aqueous Tear Deficiency; Meibomian Gland Dysfunction; Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Meibomian Gland Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study will include 30 patients enrolled in 2 stages.
  1. The first 15 patients are treated in the more severe dry eye conditioned eye.
  2. The remaining 15 patients will be treated on both eyes, applying treatment to both eyes sequentially during the same visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RMS treatment (Experimental)
  Interventions: Device: Ocular Repetitive Magnetic Stimulation (RMS) treatment

INTERVENTIONS:
Device: Ocular Repetitive Magnetic Stimulation (RMS) treatment — First stage: Patients will be asked to undergo a one-time treatment with Epitech Corneal Magnetic Stimulation Device on one eye. The worst eye will be treated; if both eyes are equal, the right eye will be treated.
  Second stage: will be treated on both eyes, applying treatment to both eyes sequentially during the same visit.

SUMMARY:
The study aims to test the safety of Repetitive Magnetic Stimulation (RMS) treatment for dry eye disease. Patients are asked to undergo a one-time treatment with Epitech Ocular Magnetic Stimulation Device on one eye in the first stage and both eyes sequentially in the second stage of the study. Changes are monitored for over a study period of 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-80 years old
2. Subjects with moderate to severe dry eye syndrome
3. Subjects able to understand the requirements of the protocol and provide informed consent.

Exclusion Criteria:

1. Eyes with other ocular surface pathology which requires more treatment than eye lubricant and conventional eyelid hygiene
2. A concurrent ocular disease including ocular infection or pterygium.
3. Ocular surgery within the previous 6 months and LASIK within the previous 1 year.
4. Any ocular injury or ocular Herpes infection within past 3 months
5. Anticipated necessity to wear contact lens in the duration of the study.
6. Unstable thyroid disorders (Drugs Tx not stable in the last 3 months).
7. Alcoholism
8. Pregnant or nursing women
9. Documented HIV positive
10. Cardiac pacemakers, cardioverter defibrillators, or neurostimulators, cochlear implants, implanted medication pumps or intracardiac lines, implanted brain electrodes (cortical or deep-brain electrodes)
11. Any Conductive, ferromagnetic or other magnetic - sensitive objects such as aneurysm clips or coils, stents, bullet fragments in the head or neck
12. Significant heart disease or cerebrovascular disease
13. History of epilepsy, dementia, head trauma, increased intracranial pressure, or central nervous system (CNS) tumors.
14. Participation in another ophthalmic clinical trial within past 30 day
15. Any other specified reason as determined by the clinical investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) | 3 mounth

CONTACTS AND LOCATIONS:
Overall Officials: Avi Solomon, MD, Principal Investigator — Hadassah Medical Organization; David Zadok, MD, Principal Investigator — Shaare Zedek Medical Center; Haggay Avizemer, MD, Principal Investigator — Wolfson Medical Center
Locations (3):
- Israel (3):
  - E. Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Center (SZMC), Jerusalem